CLINICAL TRIAL: NCT05670782
Title: A Phase 2 Study Evaluating the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of KM-819 in Healthy Older Adults and Participants with Parkinson's Disease
Brief Title: A Study to Evaluate Safety and Efficacy of KM-819 in Healthy Adults and Participants with Parkinson's Disease
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: FAScinate Therapeutics Inc. (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Organization: Kainos Medicine Inc. (Industry)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: FASCP-819-K103
Record Dates: First submitted 2022-12-21; First posted 2023-01-04 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2024-06

CONDITIONS: Parkinson Disease
Keywords: Inhibition of FAF1(Fas (TNFRSF6)-associated factor 1); Multiple Ascending Dose (MAD); Neuroprotection; Alpha-synuclein inhibition; KM-819
MeSH Terms: conditions — Parkinson Disease | interventions — KM-819

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Part 1a: Cohort 1.1a Dose 400 mg (Experimental): Healthy older adult participants will receive oral 400 mg dose of KM-819 or matching placebo once-daily for 7 days, after fasting for 2 hours prior to administration of study intervention and will be required to fast for 1 hour after administration of study intervention.
  Interventions: Drug: KM-819; Drug: Placebo
- Part 1a: Cohort 1.2a Dose 600 mg (Experimental): Healthy older adult participants will receive oral 600 mg dose of KM-819 or matching placebo once-daily for 7 days, after fasting for 2 hours prior to administration of study intervention and will be required to fast for 1 hour after administration of study intervention.
  Interventions: Drug: KM-819; Drug: Placebo
- Part 1a: Cohort 1.3a Dose 800 mg (Experimental): Healthy older adult participants will receive oral 800 mg dose of KM-819 or matching placebo once-daily for 7 days, after fasting for 2 hours prior to administration of study intervention and will be required to fast for 1 hour after administration of study intervention.
  Interventions: Drug: KM-819; Drug: Placebo
- Part 1b: Cohort 1.1b Dose 200 mg (Experimental): Participants with Parkinson's disease will receive oral 200 mg dose of KM-819 or matching placebo once-daily for 7 days, after fasting for 2 hours prior to administration of study intervention and will be required to fast for 1 hour after administration of study intervention.
  Interventions: Drug: KM-819; Drug: Placebo
- Part 1b: Cohort 1.2b Dose 400 mg (Experimental): Participants with Parkinson's disease will receive oral 400 mg dose of KM-819 or matching placebo once-daily for 7 days, after fasting for 2 hours prior to administration of study intervention and will be required to fast for 1 hour after administration of study intervention.
  Interventions: Drug: KM-819; Drug: Placebo
- Part 1b: Cohort 1.3b Dose 600 mg (Experimental): Participants with Parkinson's disease will receive oral 600 mg dose of KM-819 or matching placebo once-daily for 7 days, after fasting for 2 hours prior to administration of study intervention and will be required to fast for 1 hour after administration of study intervention.
  Interventions: Drug: KM-819; Drug: Placebo
- Part 2: Cohort 2.1 Dose X (Experimental): Participants with Parkinson's disease will receive oral doses of KM-819 (dose to be determined based on the findings from Part 1) or matching placebo once-daily for 730 days and will be allowed to take study intervention with or without fasting.
  Interventions: Drug: KM-819; Drug: Placebo
- Part 2: Cohort 2.2 Dose Y (Experimental): Participants with Parkinson's disease will receive oral doses of KM-819 (dose to be determined based on the findings from Part 1) or matching placebo once-daily for 730 days and will be allowed to take study intervention with or without fasting.
  Interventions: Drug: KM-819; Drug: Placebo

INTERVENTIONS:
Drug: KM-819 — Participants will receive oral doses of KM-819 once-daily
Drug: Placebo — Participants will receive matching placebo once-daily

SUMMARY:
The goal of this study is to test KM-819 in halting or slowing the progression of Parkinson's disease.

The study evaluates the safety and tolerability of multiple ascending doses of KM-819 in healthy older adults and participants with Parkinson's disease.

DETAILED DESCRIPTION:
The overall study will consist of three parts (Part 1a, Part 1b and Part 2).

Part 1 of this study will evaluate the safety, tolerability and plasma PK of multiple ascending doses (MAD) of KM-819 in healthy older adults (Part 1a) and participants with Parkinson's disease (Part 1b).

* Part 1a is a randomized, double-blind, Multiple Ascending Dose (MAD) study in healthy older adults that will include 3 cohorts.
* Part 1b is a randomized, double-blind, MAD study in participants with Parkinson's disease that will include 3 cohorts.

Part 2 of the study is a randomized, double-blind, multiple dose study in participants with Parkinson's disease that will include 2 cohorts. It is designed to test the safety, tolerability, plasma PK and pharmacodynamic effects of KM-819 in participants with Parkinson's disease. The study will also assess the degree to which those treated with KM-819 will experience gains in overall daily function within the context of improved Parkinson's disease motor and non-motor symptoms in comparison to placebo. Participants will be randomized to receive KM-819 or matching placebo at doses to be determined based on the findings from Part 1 in a 2:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Participant is a healthy volunteer or has a clinical diagnosis of idiopathic Parkinson's disease.
* Participant is on a stable dose of medications to treat Parkinson's disease at least 8 weeks prior to randomization
* Presence of idiopathic Parkinson's disease Hoehn and Yahr Stage ≤ 4
* History or current use of dopamine/dopaminergic drugs, levodopa with decarboxylase inhibitor or dopaminergic agonists, with a stable dosage for at least 30 days prior to Screening
* Body mass index (BMI) within the range 18.5 to 35 kg/m2 (inclusive)
* A male participant must not have a pregnant or breastfeeding partner and must agree to use a highly effective contraception method starting from Screening and refrain from donating sperm during this period
* A female participant is eligible to participate if she is not pregnant, not breastfeeding

Exclusion Criteria:

* Diagnosis of neurodegenerative disorder other than idiopathic Parkinson's disease resulting in dementia or atypical parkinsonism
* Life-time history of a suicide attempt as determined by the Columbia-Suicide Severity Rating Scale (C-SSRS) for the Screening
* Evidence of cognitive decline defined by the Montreal Cognitive Assessment (MoCA) score ≤25 for healthy normal population (Part 1a) and ≤21 for the patient population (Part 1b and Part 2)
* History of levodopa-induced motor fluctuations or dyskinesia
* Prior surgical treatment for Parkinson's disease
* Clinically significant brain abnormalities on or contraindication to a structural magnetic resonance imaging (MRI)
* Significant respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, pancreatic, musculoskeletal, genitourinary, immunological or dermatological disorders.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 314 (Estimated)
Dates: Start 2022-07-19 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-11-13 (Estimated)

PRIMARY OUTCOMES:
Part 1a,1b and 2: Number of participants with adverse events and serious adverse events | Part 1a and Part 1b: From screening (Day -42 to -3) up to 7 days and Part 2: From screening (Day -42 to -2) to 730 days
  To evaluate the safety and tolerability of multiple ascending doses of KM-819
Part 2: Change from baseline in the Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part II: Activities of Daily Living (ADL) Score at Day 730 | From screening (Day -42 to -2) to Day 730
  Activities of Daily living (ADL) will be assessed via MDS-UPDRS score. MDS-UPDRS Part II is a self-administered questionnaire that assesses the motor experience of daily living in participants with Parkinson's disease. Score: 0: Normal, 1: Slight, 2: Mild, 3: Moderate, 4: Severe. Higher the score, the more severe the condition or symptom

SECONDARY OUTCOMES:
Part 1a and 1b: Area under the concentration-time curve (AUC) from pre-dose (time zero) to the time of the last quantifiable concentration AUC(0-t) | Day 1
  To evaluate the pharmacokinetics (PK) of multiple ascending doses (MAD) of KM-819 in plasma
Part 1a and 1b: AUC from pre-dose (time zero) to 24 hours post-dose [AUC(0-24)] | Day 1
  To evaluate the pharmacokinetics (PK) of multiple ascending doses (MAD) of KM-819 in plasma
Part 1a and 1b: Maximum concentration (Cmax) | Day 1
  To evaluate the pharmacokinetics (PK) of multiple ascending doses (MAD) of KM-819 in plasma
Part 1a and 1b: Time to achieve Cmax (tmax) | Day 1
  To evaluate the pharmacokinetics (PK) of multiple ascending doses (MAD) of KM-819 in plasma
Part 1a and 1b: Minimum concentration (Cmin) | Day 1
  To evaluate the pharmacokinetics (PK) of multiple ascending doses (MAD) of KM-819 in plasma
Part 1a and 1b: AUC normalized to dose administered (AUC_D) | Day 1
  To evaluate the pharmacokinetics (PK) of multiple ascending doses (MAD) of KM-819 in plasma
Part 1a and 1b: Cmax normalized to dose administered (Cmax_D) | Day 1
  To evaluate the pharmacokinetics (PK) of multiple ascending doses (MAD) of KM-819 in plasma
Part 1a and 1b: AUC from pre-dose (time zero) extrapolated to time infinity [AUC(0-inf)] | Day 1
  To evaluate the pharmacokinetics (PK) of multiple ascending doses (MAD) of KM-819 in plasma
Part 1a and 1b: Apparent terminal elimination half-life (t½) | Day 1
  To evaluate the pharmacokinetics (PK) of multiple ascending doses (MAD) of KM-819 in plasma
Part 1a and 1b: Terminal elimination rate constant (λz) | Day 1
  To evaluate the pharmacokinetics (PK) of multiple ascending doses (MAD) of KM-819 in plasma
Part 1a and 1b: Percentage of AUCinf that is extrapolated beyond the time of the last quantifiable concentration [%AUC (extrap)] | Day 1
  To evaluate the pharmacokinetics (PK) of multiple ascending doses (MAD) of KM-819 in plasma
Part 1a and 1b: Apparent oral clearance (CL/F) | Day 1
  To evaluate the pharmacokinetics (PK) of multiple ascending doses (MAD) of KM-819 in plasma
Part 1a and 1b: AUC(0-t) at steady state (Vz/F) | Day 1
  To evaluate the pharmacokinetics (PK) of multiple ascending doses (MAD) of KM-819 in plasma
Part 1a and 1b: AUC(0-t) at steady state [AUC(0-t_ss)] | Day 7
  To evaluate the pharmacokinetics (PK) of multiple ascending doses (MAD) of KM-819 in plasma
Part 1a and 1b: AUCtau at steady state [AUC(tau_ss)] | Day 7
  To evaluate the pharmacokinetics (PK) of multiple ascending doses (MAD) of KM-819 in plasma
Part 1a and 1b: Cmax at steady state (Cmax,ss) | Day 7
  To evaluate the pharmacokinetics (PK) of multiple ascending doses (MAD) of KM-819 in plasma
Part 1a and 1b: tmax at steady state (tmax,ss) | Day 7
  To evaluate the pharmacokinetics (PK) of multiple ascending doses (MAD) of KM-819 in plasma
Part 1a and 1b: Ctrough at steady state (Ctrough_ss) | Day 7
  To evaluate the pharmacokinetics (PK) of multiple ascending doses (MAD) of KM-819 in plasma
Part 1a and 1b: Minimum concentration at steady state (Cmin,ss) | Day 7
  To evaluate the pharmacokinetics (PK) of multiple ascending doses (MAD) of KM-819 in plasma
Part 1a and 1b: Average observed concentration at steady state (Cav,ss) | Day 7
  To evaluate the pharmacokinetics (PK) of multiple ascending doses (MAD) of KM-819 in plasma
Part 1a and 1b: Accumulation ratio calculated using AUC [Rac (AUC)] | Day 7
  To evaluate the pharmacokinetics (PK) of multiple ascending doses (MAD) of KM-819 in plasma
Part 1a and 1b: Accumulation ratio calculated using Cmax [Rac (Cmax)] | Day 7
  To evaluate the pharmacokinetics (PK) of multiple ascending doses (MAD) of KM-819 in plasma
Part 1a and 1b: Apparent oral clearance at steady state (CL/Fss) | Day 7
  To evaluate the pharmacokinetics (PK) of multiple ascending doses (MAD) of KM-819 in plasma
Part 1a and 1b: AUC normalized to dose administered at steady state (AUCss_D) | Day 7
  To evaluate the pharmacokinetics (PK) of multiple ascending doses (MAD) of KM-819 in plasma
Part 1a and 1b: Cmax_ss normalized to dose administered (Cmaxss_D) | Day 7
  To evaluate the pharmacokinetics (PK) of multiple ascending doses (MAD) of KM-819 in plasma
Part 1a and 1b: Fraction of dose excreted in urine (Fe) | Day 7
  To evaluate the pharmacokinetics (PK) of multiple ascending doses (MAD) of KM-819 in urine
Part 1a and 1b: Renal clearance (CLR) | Day 7
  To evaluate the pharmacokinetics (PK) of multiple ascending doses (MAD) of KM-819 in urine
Part 2: Sparse plasma PK blood sampling for population PK analysis | Day 1, Day 7, Day 30 and Day 180
  Sparse plasma population PK sampling will be collected, and population PK modeling will be used to characterize the PK of KM-819 in participants with Parkinson's disease.

OTHER OUTCOMES:
Digital biomarkers using the Parkinson's Disease Digital Biomarker Solutions from Roche Molecular Solutions. | From screening (Day -42 to -2) to 2 years
  Measurements of active and passive monitoring of Parkinson's disease symptoms utilizing smartphone based devices and software

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Parexel Early Phase Clinical Unit, Glendale, California
  - University California San Diego Medical Center, San Diego, California
  - Quest Research Institute, Rose Cancer Center, Royal Oak, Michigan

IPD SHARING:
Plan to Share IPD: Undecided
Individual Identifiable personal information will not be shared. All individuals will be coded.